CLINICAL TRIAL: NCT01493271
Title: An Adaptive, Multi-center, Randomized, Investigator-masked, Subject-masked, Multiple-dose, Placebo-controlled, Parallel Study to Investigate Efficacy, Safety, Tolerability and Pharmacokinetics of RO5093151 for up to 28 Days in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension.
Brief Title: A Study of RO5093151 in Patients With Ocular Hypertension Or Open Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP25466
Record Dates: First submitted 2011-12-14; First posted 2011-12-15 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension, Glaucoma, Open-Angle
MeSH Terms: conditions — Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO5093151 (Experimental)
  Interventions: Drug: RO5093151

INTERVENTIONS:
Drug: Placebo — Placebo to RO5093151
  Arms: Placebo
Drug: RO5093151 — oral doses twice daily for up to 28 days
  Arms: RO5093151

SUMMARY:
This randomized, double-blind, placebo-controlled, multi-center study will evaluate the safety and the effect of RO5093151 on intraocular pressure in patients with ocular hypertension or open angle glaucoma. Patients will be randomized to receive oral doses of RO5093151 or placebo twice daily. The anticipated time on study treatment is 7 days with the possibility to extend to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, at least 21 years of age, inclusive
* Diagnosis of ocular hypertension or primary open angle glaucoma in at least one eye
* Able to participate and willing to give informed consent

Exclusion Criteria:

* Presence of extreme narrow angle with complete or partial closure
* Progressive retinal or optic nerve disease from any cause other than glaucoma
* History or signs of penetrating ocular trauma
* Uncontrolled hypertension
* Clinically significant abnormalities in laboratory test results
* Positive test results on hepatitis B, hepatitis C, or HIV 1 and 2
* Kidney disease or dysfunction

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in mean intraocular pressure (IOP) at 1 hour post-dose following 7 days of treatment | Day 7

SECONDARY OUTCOMES:
Change in mean daily intraocular pressure (IOP) | Up to 28 days
Change in mean intraocular pressure (IOP) at each assessment time-points | Up to 28 days
Change in intraocular pressure (IOP) during a placebo lead-in phase | 7 days
Pharmacokinetics (area under the concentration time curve) | Day 7
Urinary ratio of tetrahydrocortisol to tetrahydrocortisone | 7 days
Safety (incidence of adverse events) | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- United States (3):
  - Morrow, Georgia
  - High Point, North Carolina
  - Mt. Pleasant, South Carolina
- Sofia, Bulgaria
- Czechia (5):
  - Hradec Králové
  - Litomysi
  - Prague
  - Ústí nad Labem
  - Zlín
- Hungary (2):
  - Budapest
  - Esztergom